CLINICAL TRIAL: NCT06796959
Title: Combined [18F]-FDG PET-MRI in Diagnostics and Surveillance of Small Bowel Crohn's Disease (CD-PET)
Brief Title: Combined [18F]-FDG PET-MRI in Diagnostics and Surveillance of Small Bowel Crohn's Disease
Acronym: CD-PET
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Finnish governmental support for health sciences (Unknown); Mary and Georg Ehrnroot's foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: ETMK 49/2019
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Small Bowel Crohn's Disease
Keywords: small bowel Crohn's disease; ileitis
MeSH Terms: conditions — Ileitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Tissue samples from small bowel Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study subjects: Patients with suspected small bowel Crohn's disease

SUMMARY:
Patients with suspected small bowel Crohn's disease (CD) are assessed with PET-MRE using 18-fluorodeoxyglucose ([18F]-FDG) tracer. Patients are recruited from the outpatient clinic of gastroenterology in Turku University Hospital. The patients must fulfil the eligibility criteria and give their signed approvement prior to their enrolment into the study. This is an observational single-center imaging study.

35 patients with high clinical suspicion of active small bowel CD will be enrolled to study. After the diagnostic [18F]-FDG-PET-MRE, patients will undergo small bowel capsule endoscopy (SBCE) if no strictures are seen in PET-MRE. [18F]-FDG-PET-MRE will be repeated in 3 months after medical therapy for CD has been started. Medical therapy will be started by clinicians blinded from PET-data but have access to MRE-data and all other diagnostic measures. Adequate medication is chosen by clinicians not participating in the study and thus enrollment does not affect the choice of medical therapy for patients participating in this study. [18F]-FDG-PET-MRE and clinical assessment of disease activity will be performed within 1 month of recruitment. Follow up-visits will be arranged in the outpatient clinic of gastroenterology in Turku University Hospital.

The aim is to investigate whether [18F]-FDG-PET-MRE can be used in diagnostics and follow-up of small bowel CD and to compare its performance to MRE.

DETAILED DESCRIPTION:
Diagnostics and follow up of small bowel CD can be difficult, large parts of small bowel can't be assessed by conventional endoscopy. MRE can detect transmural lesions, but sensitivity is limited with luminal disease. SBCE can detect even small lesions, but specificity is low. More accurate tools for diagnostics are hence needed. Our aim is to is to show that [18F]-FDG-PET-MRE can be used in diagnostics and disease activity monitoring of small bowel CD

Volunteer patients with clinically suspected small bowel CD (i.e. ileitis in colonoscopy, diarrhea, anemia and elevated fecal calprotectin or suspected CD in cross sectional imaging) are recruited from the outpatient clinic of gastroenterology in Turku University Hospital. The patients must fulfil the eligibility criteria and give their signed approvement prior to their enrolment into the study. All patients have previously been in ileocolonoscopy.

After screening, the patients have routine blood samples taken. A complete blood count (CBC), C-reactive protein (CRP), creatinine, alanine aminotransferase (ALAT), alkaline phosphatase (AFOS) and albumin will be analyzed from each patient's blood sample and fecal calprotectin analyzed from stool. Patients are then assessed with PET-MRE using 18-fluorodeoxyglucose ([18F]-FDG) tracer. The patients must fulfil the eligibility criteria and give their signed approvement prior to their enrolment into the study.

Patients fast for six hours prior to PET-MRE study. Oral mannitol is used as enteral contrast. Venous catheters will be placed at both antecubital veins for injection of [18F]-FDG and gadolinium contrast agent for MRE-sequences. Patients will lie prone for approximately 1.5h during the PET-MRE imaging. Prior to imaging, fasting glucose is measured from venous blood. During the imaging, FDG -activity will be measured from venous blood. The uptake of FDG in small bowel will be measured from the images obtained from segments with inflammation and healthy-looking segments for comparison.

If no strictures are present in the PET-MRE, the patients will go through SBCE to confirm the diagnosis of small bowel CD. The patients are arranged a visit to clinician in the outpatient clinic of gastroentereology in Turku University Hospital. The clinicians have access to MRE-data, endoscopy and SBCE-data and laboratory data, but are blinded from PET-results to avoid bias. The clinicians choose adequate treatment for each patient individually following general guidelines (such as ECCO) of treatment of small bowel CD. The patients diagnosed with small bowel CD will undergo a repeated PET-MRE following the same protocol as the first diagnostic PET-MRE to assess response to therapy. After the follow-up PET-MRE, patients medical history including laboratory and medication data will be followed and gathered for 12 months.

Primary outcome is to show that standardized uptake values (SUV) measured in [18F]-FDG-PET-MRE are higher in patients with CD than in patients not diagnosed with CD.

Secondary outcome is to show that starting effective medical therapy to small bowel CD decreases SUV in small bowel segments with CD inflammation. Secondary aim is also to investigate whether changes in SUV can predict long term disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* clinically suspected small bowel CD
* or ileitis in colonoscopy
* or diarrhea or anemia and elevated fecal calprotectin
* or suspected CD in cross sectional imaging)

Exclusion Criteria:

* age under 18 or above 70
* pregnancy
* metformin-medication
* claustrophobia
* previously known small bowel CD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled from outpatient clinic of gastroenterology of Turku University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Standard uptake value in diagnostics of small bowel CD | Immediate
  Primary outcome is to show that standard uptake values (SUV) measured in [18F]-FDG-PET-MRE are higher in patients with CD than in patients not diagnosed with CD.

SECONDARY OUTCOMES:
Change in standardized uptake values (SUV) in follow-up | Six months
  Secondary outcome is to show that starting effective medical therapy to small bowel CD decreases SUV in small bowel segments with CD inflammation. Secondary aim is also to investigate whether changes in SUV can predict long term disease outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku PET Center, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Study data were collected from Turku University Hospital electronic patient database. Anonymized research data sets will be preserved and made accessible through the Finnish Social Science Data Archives once the whole project is finalized. Further inquiries can be directed to the primary investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1.8.2020-1.8.2030
Access Criteria: Anonymized research data sets will be preserved and made accessible through the Finnish Social Science Data Archives once the whole project is finalized.

REFERENCES:
- [Background] Mattila J, Kallio J, Loyttyniemi E, Nuutila P, Koffert J. Combined [18F]-Fluorodeoxyglucose Positron Emission Tomography-MR Imaging: A Promising Tool for Diagnostics of Small Bowel Crohn's Disease. Dig Dis. 2025;43(1):104-114. doi: 10.1159/000542379. Epub 2024 Nov 13. PMID 39536721
- [Derived] Mattila J, Kallio J, Loyttyniemi E, Nuutila P, Koffert J. Combined [18F]-FDG PET-MR imaging for monitoring small bowel crohn's disease. Eur J Nucl Med Mol Imaging. 2026 Jan;53(2):1234-1245. doi: 10.1007/s00259-025-07524-4. Epub 2025 Aug 26. PMID 40856818